CLINICAL TRIAL: NCT04498377
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Multicenter Study to Evaluate the Efficacy and Safety of F-652 (IL-22:IgG2 Fusion Protein) in Patients With Moderate to Severe COVID-19
Brief Title: Study of F-652 (IL-22:IgG2 Fusion Protein) in Patients With Moderate to Severe COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There have been significant changes in the FDA guidelines and clinical standard of care
Sponsor: EVIVE Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC-652-04
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — eflepedocokin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized in a 1:1 ratio in a double-blind manner to receive F-652 or placebo.
  An independent statistician from Medpace will generate the randomization schedule. Patients meeting eligibility criteria will be randomized on Day 1 in a 1:1 ratio to F-652 or placebo, respectively. Patients will be assigned a randomization number and treatment assignment according to the randomization schedule. This randomization schedule will be maintained by the investigative site pharmacist until it is appropriate to break the blind. The Investigator, investigative site personnel (except site-designated pharmacist and dedicated assistant), study monitors, vendors, Sponsor, and Medpace will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- F-652 (Experimental): Patient receives standard care plus F-652
  Interventions: Biological: F-652
- Placebo (Placebo Comparator): Patient receives standard care plus placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: F-652 — IL-22 fusion protein administered intravenously
  Arms: F-652
Biological: Placebo — Placebo administered intravenously
  Arms: Placebo

SUMMARY:
This is an interventional, multicenter, 2-arm, parallel-group, randomized, double-blind, placebo controlled, dose-escalation, safety and efficacy study of F-652 treatment versus placebo in patients aged 18 years or older with a COVID-19 diagnosis confirmed by PCR. Eligible patients will have moderate to severe COVID-19 symptoms within 5 days post hospitalization and a positive COVID-19 testing.

DETAILED DESCRIPTION:
The study is planned to include 4 cohorts, with enrolled patients being randomized 1:1 in a blinded manner on Day 1, following screening, to F-652 or placebo as follows:

* Cohort 1 (sentinel cohort): Four patients will receive either dose level 1 F-652 or placebo. Upon completion of sentinel, the Data Monitoring Committee will evaluate the safety and tolerability data of the sentinel patients and determine if it is acceptable to dose the remaining patients in this dosing group in Cohort 2.
* Cohort 2: Fourteen patients will receive either dose level 1 F-652 or placebo. Upon completion of Cohort 2, the DMC will convene and review all available safety data to determine if the study can proceed to the next dose level.
* Cohort 3 (sentinel cohort): Four patients will receive either dose level 2 F-652 or placebo. Upon completion of sentinel dosing, the DMC will evaluate the safety and tolerability data of the sentinel patients and determine if it is acceptable to dose the remaining patients in this dosing group in Cohort 4.
* Cohort 4: Sixteen patients will receive either dose level 2 F-652 or placebo. Treatment will begin on Day 1 following randomization. Patients assigned to active drug will receive a total of 2 doses of F-652 (1 IV infusion on Day 1 and 1 IV infusion on Day 8). Patients assigned to placebo will receive identical IV infusions of placebo vehicle on Days 1 and 8. All patients will receive available supportive and antiviral therapies as standard of care. Efficacy will be assessed on Days 15 and 29. Patients will be followed for safety until Day 60.

The primary efficacy endpoint is the proportion of patients with a ≥2-point increase in the National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale from baseline to Day 29.

The secondary efficacy endpoints include the proportion of patients with a ≥2-point increase in the NIAID 8-point ordinal scale from baseline to Day 15, mortality rate by Days 15 and 29, percentage of patients who have recovered and discharged from the hospital by Days 15 and 29, and percentage of patients progressed to severe/critical disease by Day 15.

The safety endpoints include all cause treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs); change from screening (baseline) in clinical symptoms and abnormal vital signs, abnormal laboratory tests; and relationship of any AEs with F-652 treatment.

The exploratory endpoints include time to negative SARS-CoV-2 PCR test from randomization; and changes in pharmacodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent and able to comply with protocol requirements
* 18 years or older
* Has a COVID-19 diagnosis confirmed by PCR
* Hospitalized within 5 days and meets the following criteria at screening:

Peripheral capillary oxygen saturation (SpO2) ≤ 93% on room air or SpO2 ≥93% on ≤10 liters per minute of supplemental oxygen via nasal cannula

* Radiographic (chest X-ray, computed tomography scan, or ultrasound) evidence of bilateral pulmonary infiltrates consistent with SARS-CoV-2/COVID-19
* Clinical symptoms consistent with COVID-19 per Investigator judgement
* Body mass index between 18 to 40 kg/m2
* If of reproductive potential, willing to abstain or agree to the use of highly effective contraception

Exclusion Criteria:

* Respiratory failure at screening
* History of heart failure
* History of COPD or bronchial asthma
* Active TB or history of TB of the following types
* Uncontrolled arrhythmia within 3 months prior to randomization
* Heart disease of the following types
* Moderate to severe renal insufficiency
* Abnormal white cell and platelet counts
* History of transplantation of vital organs (e.g., heart, lung, liver, and/or kidney);
* Malignant tumor
* Uncontrolled systemic or local autoimmune or inflammatory disease besides SARS-CoV-2
* Unhealed wounds, active gastric ulcer, had surgery
* Received other investigational therapeutic products
* Used interferon therapies
* History of HIV infection, hepatitis B, and/or hepatitis C
* Known serious allergic reaction or hypersensitivity to components of F-652
* Pregnant or breastfeeding
* History of drug abuse or use of narcotics
* Treated with immunomodulators or immunosuppressants
* Other conditions resulting in increased risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Bojanowski, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | F-652 | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study enrolled only 1 patient in F-652 arm, no patient enrolled in placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | F-652 | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: NIAID 8-point Ordinal Scale
Description: The proportion of patients with a greater or equal 2-point change in the National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale from baseline to Day 29.
  The NIAID 8-point ordinal scale includes the following grades:
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation;
  3. Hospitalized, on non-invasive ventilation or high-flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplementation oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  7. Not hospitalized, limitation on activities and/or requiring home oxygen; and
  8. Not hospitalized, no limitations on activities.
Time Frame: Study day 1 before dose to day 29
Population: Only 1 patient enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | F-652 | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Description: There is 1 patient enrolled in F-652 arm, no patient enrolled in placebo arm.
Arm/Group | F-652 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-652 (N=1) | Placebo (N=0)
Chills (General disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT04498377/Prot_SAP_001.pdf